CLINICAL TRIAL: NCT04883463
Title: Neuromodulation to Improve Respiratory Function in Cervical Spinal Cord Injury
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Daniel Lu, MD, PhD, Associate Professor of Neurosurgery, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-000994; UH3NS119772 (NIH)
Record Dates: First submitted 2020-11-24; First posted 2021-05-12 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: Spinal Cord Injuries
Keywords: Neuromodulation; Respiratory SCI; Implant
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Epidural Stimulation for Respiratory Function (Experimental): Self-controlled longitudinal safety and feasibility of stimulation and respiratory training.
  Interventions: Device: Epidural stimulation

INTERVENTIONS:
Device: Epidural stimulation — Epidural electrical stimulation implant weekly sessions for 21 months.

SUMMARY:
This is a phase 1 study of safety and feasibility of cervical spinal cord stimulator implantation in cervical SCI subjects who are ventilator dependent. The Investigators will be focusing on the safety and feasibility of this approach. Participants may qualify for the study if they are male or female 18-75 years old, are at least 1 year after original injury, have injury at C2 to C7 level, and dependent on mechanical ventilation to help them breathe. Additionally, they need to be able to attend up to twice weekly testing sessions for up to 21 months.

DETAILED DESCRIPTION:
There are five main phases to this study. The first phase is baseline testing, second phase is temporary implant, third phase is post-temporary implant mapping/treatment, fourth phase is permanent implant, and fifth phase is post-permanent implant treatment.

Phase 1. Screening and Baseline testing/training (up to 6 months, UCLA Semel Institute for Neuroscience and Human Behavior), the purpose of which is to ensure that each subject begins with the full benefits achievable by standard rehabilitative respiratory therapy and has stable baseline of function before they begin epidural stimulation. 12 subjects will undergo this phase. Maximum inspiratory and expiratory pressure, resting spontaneous respiratory activity, and respiratory muscle EMG will be measured during this phase. Subjects on ventilator assist mode (unless or until they can sustain adequate respiration on their own) will be monitored via pneumotachometer for respiratory frequency changes. Additionally, subjects will undergo motor and sensory testing. The subjects must show stable respiratory function before implantation, therefore if a subject is showing small improvements at 3 months the subject will continue training until they have reached their maximal effect from training (up to 6 months). Subjects that show stable baseline at 3 months will proceed to Phase 2. If a subject's health worsens, including non-respiratory functioning, subject will be assessed by appropriate physician and testing will be held until subject's health has improved and maintains stable for at least 2 months. Subjects will obtain preoperative clearance and general anesthesia clearance in preparation for Phase 2.

Phase 2. Temporary Implant (1 day, 24 hours overnight stay, UCLA Medical Center, Santa Monica). Subjects will undergo temporary stimulator implant surgery. CT scan may be collected prior for surgical planning if needed by PI. Up to 9 subjects with most connectivity and evidence of response to baseline testing will undergo this phase from the pool of 12 subjects in Phase 1 above. The electrode that will be used will be the same one that will be applied in subsequent permanent trial Phase 4, however a temporary connector will be placed to an external battery source and no permanent battery will be implanted. Connectivity of subject will be based on motor evoked potentials and somatosensory evoked potentials done during baseline testing and evaluated by a clinical neurophysiologist

Phase 3. Post-temporary implant mapping/treatment. Respiratory ability will be assessed. Respiratory rehabilitation regimen with the stimulator will be used to re-enable respiratory function. The length of time of this phase will be dependent on the participant's response (as explained below) to the implant. The paddle will remain implanted until a comprehensive assessment of the participant's respiratory response is conducted by PI. Should the participant fail to exhibit a measurable respiratory response, the explantation of the paddle electrodes may be performed by the PI, provided that it is deemed safe to proceed. Extent and amplitude of evoked responses and motor pools activated from electrode pairs will be analyzed through EMG obtained. Response to the temporary stimulator implant will be based on tidal volume and spontaneous respiratory rate and respiratory muscle EMG. The same 9 subjects from Phase 2 will undergo this phase. Maximum inspiratory and expiratory pressure, and respiratory muscle EMG measurements will also be collected during this Phase.

Phase 4. Permanent implant procedure (1 day, 24 hours overnight stay, UCLA Medical Center, Santa Monica). Subjects will undergo stimulator implant surgery. Up to 6 subjects with most connectivity and evidence of response to baseline testing will undergo this phase from the pool of 9 subjects in Phase 3 above. The functional respiratory circuit connectivity of the subject will be based on implanted spinal cord stimulator-induced spinal evoked respiratory muscle potential changes. Response to stimulator implant-induced respiratory facilitation will be evaluated based on intraoperative minute ventilation, tidal volume, and respiratory muscle EMG before and after the spinal stimulation. Subjects will be monitored overnight following surgery as a pre-cautionary measure. Ventilated subjects undergoing surgery are not at an increased risk over non-ventilated subjects.

Phase 5. Post-permanent implant mapping/treatment (up to 12 months, UCLA Semel Institute for Neuroscience and Human Behavior) in which the electrode pair or pairs that maximally activate the largest number of respiratory motor pools will be identified based on the extent and amplitude of evoked responses in the respiratory muscles. Connectivity of subject will be based on motor evoked potentials and somatosensory evoked potentials done during baseline testing and evaluated by a clinical neurophysiologist. Response to respiratory training will be evaluated based on pulmonary function tests (including tidal volume, maximum inspiratory and expiratory effort, spontaneous respiratory activity) and respiratory muscle EMG. Once optimal parameters have been identified, electrode pairs that allow subjects to manipulate their respiratory frequency with concomitant diaphragm/intercostal EMG activity, subjects will be allowed to use stimulator at home (daily, with identified parameters) with respiratory training in addition to weekly (or monthly) testing. Each subject will undergo stimulation up to twice a week in the clinic and daily (with identified parameters) up to 12 months. Extent and amplitude of evoked responses and motor pools activated from electrode pairs will be analyzed through EMG. Respiratory rehabilitation regimen with the stimulator will be used to re-enable respiratory function. 6 subjects will be tested up to twice weekly in the clinic for up to 2 hours per session. Pulmonary function tests (including maximum inspiratory and expiratory pressure, resting spontaneous pressure, and initiated breaths) will be evaluated weekly or monthly. Post-implant MEP/SSEP, SCIM3, FIM, ISNCSCI, SCI-QOL testing will be conducted at a minimum of one timepoint during this phase of the study. For patients with a ventilator, home use will involve turning on the stimulator, breathing with the ventilator, and turning the sensitivity of ventilator assist mode up, working to strengthen the muscles for initiated breaths. The same 6 subjects from Phase 4 will undergo this phase.

Timeline. The study is a safety and feasibility trial. This is a single arm implantation of permanent electrode to assess safety and early efficacy of cervical spinal epidural stimulation to improve respiratory function. It is conducted over a period of up to 6 months or 21 months in 1, 2, or 3 periods, respectively: Phase 1. Baseline training (up to 6 months), Phase 2. Temporary Trial Implant (1 day), Phase 3. Post-temporary trial implant treatment (the length of time of this phase will be dependent on participant's response to the implant), Phase 4. Permanent Implant (1 day, with up to 2 months for surgical recovery), Phase 5. Post-permanent implant treatment (up to 12 months). Therefore, 12 subjects will be involved for up to 6 months, while 9 subjects will be involved for up to 7 months, and 6 subjects involved for up to 21 months (18 months of testing with up to 2 months recovery).

Home Use. To ensure safety, the ventilator will provide support for the patient during home use with stimulator turned on, just as it does when epidural stimulation is not on. The patient will not be completely disconnected to the ventilator unless independence from the ventilator is achieved through a gradual and very closely supervised weaning process in which the patient will demonstrate stable O2 saturation and adequate minute ventilation through the stages of weaning. Weaning (and evidence of improved respiratory muscle function) will consist of gradually reducing the level of support delivered by the ventilator while requiring that as weaning occurs, the patient maintains stable minute ventilation on his own.

To ensure safety, these weaning maneuvers will be conducted only with respiratory therapist being present, and an AMBU bag with supplemental O2 will be available. Additionally, for safety, the caregiver will obtain heart rate, blood pressure, temperature at 15 min intervals and O2 saturation continuously, or when there is a change in the ventilator setting. Additionally this will be performed only when the subject is fully conscious, awake, and following commands.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 18-75 years
2. At least 1 year from initial cervical spinal cord injury
3. Non-progressive Spinal Cord Injury (SCI) at C2 - C7 (non-conus injury)
4. Motor Complete ASIA Impairment Scale (A, B, or C)
5. Severe respiratory function compromise requiring dependency on invasive or noninvasive ventilation
6. Able to attend weekly testing sessions for up to 21 months.
7. Have intact chest/lung, upper and lower extremity anatomy. The neuromuscular connections between the spinal cord and its effector muscles (respiratory and extremity) are required to be intact
8. Have intact cognitive ability, able to follow commands/voice concerns, and give consent

Exclusion Criteria:

1. History of severe autonomic dysreflexia
2. Phrenic nerve or diaphragm pacer
3. Phrenic nerve paralysis
4. Musculoskeletal dysfunction, unhealed fracture, pressure ulcer of grade 3 and above in the European Pressure Ulcer Advisory Panel Grading System, active infection
5. Clinically significant depression or ongoing drug abuse as documented in the medical record
6. Received lung surgery within one year prior to study enrollment or has active intrinsic lung disease (e.g. COPD, acute or chronic lung infection, moderate to severe asthma, emphysema, cystic fibrosis, etc.)
7. Cardiopulmonary disease that precludes training or rehabilitation
8. Other implanted stimulation devices
9. Pregnant
10. Severe cardiac disease (e.g. heart failure, atherosclerosis, arrhythmia, stroke, etc.)
11. Subjects involved in other clinical trials not associated with this trial
12. Botox injections in respiratory associated muscles within the last 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-09-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4 | 2.5 years
  International Standards for Neurological Classification of Spinal Cord Injury/American Spinal Injury Association (ISNCSCI/ASIA)- Neurological motor and sensory function given a score A-E: Timeframe: completed at the beginning and end of the phases.
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4 | 2.5 years
  Resting Spontaneous Respiratory Activity (measured in Breathes per Minute), Maximal Inspiratory Pressure (measured in cmH2O) and Spinal Cord Independence Measure (a score from 0-100) questionnaire: Timeframe: assessed weekly through the duration of the study. Data will be analyzed to compare each individual's function to their own at the beginning of the study, during the baseline period.
Incidence of Treatment-Emergent Adverse Events as assessed by CTCAE v4 | 2.5 years
  Blood Pressure (mm/Hg): Timeframe: completed at the beginning and end of each testing session.

SECONDARY OUTCOMES:
Evaluating Pulmonary Function Throughout the Duration of the Study; 20% increase in minute ventilation. | 2.5 years
  Tidal Volume = mL Timeframe: assessed weekly through the duration of the study.
Evaluating Pulmonary Function Throughout the Duration of the Study; 20% increase in minute ventilation. | 2.5 years
  Maximal Expiratory Pressure = cmH2O Timeframe: assessed weekly through the duration of the study.
Evaluating Pulmonary Function Throughout the Duration of the Study; 20% | 2.5 years
  Functional Residual Capacity = mL/kg Timeframe: assessed weekly through the duration of the study.
Evaluating Pulmonary Function Throughout the Duration of the Study; 20% | 2.5 years
  Peak Expiratory Flow Rate = mL/min Timeframe: assessed weekly through the duration of the study.
Evaluating Pulmonary Function Throughout the Duration of the Study; 20% | 2.5 years
  Minute Volume (measured in L/min): Timeframe: assessed weekly through the duration of the study. Data for all of the assessments mentioned above will be analyzed to compare each individual's function to their own at the beginning of the study, during the baseline period.Electromyography (EMG): Respiratory muscle activity will be assessed with common practice EMG recording and functional measurements. Timeframe: assessed weekly through the duration of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C Lu, MD, PhD, Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - Semel Institute of Neuroscience at UCLA, Los Angeles, California
  - UCLA Clinical and Translational Research Center, Los Angeles, California